# **Title:** Pragmatic Cyclical Lower Extremity Exercise Trial for Parkinson's disease

**NCT#:** NCT04000360

**Document Date:** 12/28/2021

Master Informed Consent Version: 9/21/2021 Site Specific Information Version: 9/24/2019

# Consent to Participate in a Research Study

PART 1: Master Consent

Study title: Pragmatic Cyclical Lower Extremity Exercise for Parkinson's Trial

**Sponsor: NIH** 

Funding Source: National Institute of Health

Grant Principal Investigator: Dr. Jay L. Alberts, PhD

You are being invited to take part in a research study. This study is a multi-site study, meaning it will take place at several different locations. Because this is a multi-site study this consent form includes two parts. Part 1 of this consent form is the Master Consent and includes information that applies to all study sites. Part 2 of the consent form is the Study Site Information and includes information specific to the study site where you are being asked to enroll. Both parts together are the legal consent form and must be provided to you.

#### Please note:

- You are being asked to participate in a research study
- Ask as many questions as needed so you can make an informed decision.
- Carefully consider the risks, benefits, and alternatives of the research.
- Your decision to participate is completely voluntary and will have no effect on the quality
  of your medical care if you choose not to participate. You can also withdraw from the study
  at any time.

#### KEY INFORMATION

The following is a short summary of this research study to help you decide whether or not to be a part of this research study. More detailed information is included later on in this document.

#### What is the purpose, procedures and duration of this study?

You are being asked to participate in this research because you have Parkinson's disease. This study is being conducted to gather information regarding the effects of a home exercise stationary cycling program on the symptoms of Parkinson's disease.

If you participate in this research, you will be randomized into one of two groups: a Usual Care group (no exercise through the research) or an Exercise Group.

Please note: To participate in this study, you must have Wi-Fi (wireless internet) in your home, and a smartphone.

Your participation in the research will last about 12 months, with assessments at baseline, and every 6 months after that.

Approval Date: 12/28/2021 Expiration Date: 12/27/2022


More detailed information can be found under the section labeled: "Information on the Research."

#### Why might you choose not to participate in this research study?

You may not want to participate in the research if you do not wish to exercise on a bicycle, or do not have home Wi-Fi or a smartphone. You may feel uncomfortable when you are asked to withhold your Parkinson's disease medication.

More detailed information about the risks of this study can be found in the section labeled "Risks."

#### Why might you choose to volunteer for this research study?

You may or may not benefit from participating in this study. Taking part in this study will help researchers learn the impact of an exercise program on the symptoms of Parkinson's disease.

More detailed information about the risks of this study can be found in the section labeled "Benefits."

### What are my other choices if I do not take part in this study?

The alternative to being in this study is to not take part.

More detailed information about the alternatives to this study can be found in the section labeled "Alternatives."

#### **DETAILED INFORMATION**

The following is more detailed information about this study in addition to the information listed above.

## INFORMATION ON THE RESEARCH

#### Why is the research study being done?

You are being asked to participate in this research because you have Parkinson's disease. This study is being conducted to gather information regarding the effects of a home exercise stationary cycling program on the symptoms of Parkinson's disease.


#### How Many People Will Take Part in this Study?

Approximately 250 individuals will participate in this research, either through the Cleveland Clinic main campus (Cleveland, Ohio), or the University of Utah (Salt Lake City, Utah). This study is being funded by a grant from the National Institute of Health (NIH).

#### What is involved if you decide to take part in this research study?

If you participate in this research, you will be randomized into one of two groups: a Usual Care group (no exercise through the research) or an Exercise Group.

*Please note:* To participate in this study, you must have Wi-Fi (wireless internet) in your home, and a smartphone. These two items are necessary to utilize the cycling platform and the activity monitor required for participation. These items are not financially covered through the research.

#### Telephone Exercise Screening:

• A member from the research team will ask you questions from the American College of Sports Medicine (ACSM) Pre-participation Health Screen to determine if it is safe for you to enter into an exercise study. If the ACSM screen recommends you acquire medical clearance, you must obtain this through your health care provider prior to study enrollment. This will not be financially covered through the research. You may not enroll into the study without either clearing the health screen or receiving medical clearance.

# Baseline Assessments (Please see Task Table Below for a List of Assessment Dețails-Assessments last Approximately 60 Minutes):

- Day 1: You will arrive for your appointment on your regular Parkinson's disease medications. You will complete the informed consent process, complete quality of life questionnaires, and be randomized for the order of your next two baseline appointments (on and off PD meds, see below), and to which study group you will take part in (Peloton or Usual Care Group- see below).
- Days 2 and 3 (on and off PD meds-order randomized): You will complete a clinical assessment, assessments on an iPad, a walking assessment, and a balance assessment.

"Off" Parkinson's disease Medication Appointment: You will be asked to refrain from taking your Parkinson's disease medications for 12 hours prior to your appointment. You should still take all of your medications for other conditions. Please bring your Parkinson's disease medications with you; you may take them immediately after your assessments.


"On" Parkinson's disease Medication Appointment: Please take your closest dose of Parkinson's disease medications one hour before your clinical testing appointment.

#### **Group Randomization:**

- All participants will be randomized into their study group during their first baseline appointment
- You will be randomized into either the Usual Care group, or the Exercise Group
- You do not have a choice regarding which group you enter

#### Research Equipment and its Usage:

This study involves the usage of a Garmin activity monitor for all participants, and
a Peloton bicycle for Exercise participants. There is no cost associated to you for
any equipment, its usage, its delivery, or its pick-up.

#### **Usual Care Group Activities:**

- You will be given a Garmin activity monitor to wear. You will also be asked to
  download the Garmin application onto your smartphone. Research personnel will
  be able to view your daily physical activity through Garmin's on-line portal. Only a
  study number will identify you through this portal. You may keep the Garmin
  activity monitor at the conclusion of the study.
- You will receive bi-weekly telephone calls from research personnel. During these
  calls, you will be asked to report any falls (if applicable). Research personnel will
  also review your Garmin activity.
- You will be asked to complete additional clinical assessments every 6 months post baseline: 6 months (off PD meds), and 12 months (off PD meds) (please see timeline diagram below)

#### **Exercise Group Activities:**

- You will be given a Garmin activity monitor to wear. You will also be asked to
  download the Garmin application onto your smartphone. Research personnel will
  be able to view your daily physical activity through Garmin's on-line portal. Only a
  study number will identify you on this portal. You may keep the Garmin activity
  monitor at the conclusion of the study.
- You will schedule a time for a Peloton bicycle to be delivered to your home at a
  time that is convenient to you. There is no cost to you for the bicycle or its delivery
  before or after the study. The company that delivers the bicycle will be contracted
  through the research staff to deliver the bicycle at the beginning of the study, and


pick up the bicycle at the conclusion of the study at a convenient time to you. The Peloton delivery technician will also set your bike to the seat settings that were determined to be best for you at your baseline appointment.

- You will be asked to cycle 3 times per week for 12 months with recommendations from research personnel
- You will receive bi-weekly telephone calls from research personnel. During these
  calls, you will be asked to report any falls (if applicable). Research personnel will
  also review your Peloton and Garmin activity. You will be asked to complete
  additional clinical assessments every 6 months post baseline: 6 months (off PD
  meds), and 12 months (off PD meds) (please see timeline diagram below)

#### Study Flow/Timeline Diagram

| | | Baseline Clinical Assessments (three total) | |
|---|---|---|---|
| Enrollment | | Randomization | |
| | Bike Fitting (after randomization) | | |
| Exercise<br>Initiation | Home Exercise<br>(125 people) | | Usual Care<br>(125 people) |
| <b>\</b> | Peloton Bike Delivery & Fitting: Begin Cycling Protocol 3 times per week | | |
| 6 months<br>↓ | Assessment<br>(off PD meds) | 3 | Assessment<br>(off PD meds) |
| | Cycling 3 times per<br>week on the<br>Peloton cycle | | |
| 12 months<br>(End of<br>Research<br>Participation) | Assessment<br>(off PD meds) | | Assessment<br>(off PD meds) |

## Assessment Details: (Baseline, +6 months, and +12 months)

| Task: | rmed Please ask any questions you may have. |
|---|---|
| Informed<br>Consent<br>Interview: | |
| Quality of Life<br>Questionnaires: | You will be asked to complete quality of life questionnaires related to your Parkinson's disease. |
| Clinical Testing: | Unified Parkinson's Disease Rating Scale Assessment: This is the same test you likely complete as standard of care by your neurologist, and involves items such as tapping your fingers and toes, standing up from a chair, and walking while a clinical specialist monitors and rates your movements. |
| iPad<br>Assessments: | Tusic 2 destriptions: |
| Six Minute<br>Walk Test: | As a measure of cardiovascular fitness, you will be asked to walk for six continuous minutes. At the conclusion of six minutes, the distance you walked, heart rate, and oxygen saturation will be recorded. *All assessments are non-invasive. |

#### Fall Questionnaire (Completed at Home)

You will be given a binder with instructions on how to record near falls and falls on papers in the binder, if applicable. You will fill this out through the entire course of the study duration (12 months), regardless of whether or not you experienced a fall during the week. You will be asked to have your binder with you during the study bi-weekly telephone calls.

#### How will my data be used?

If you choose to participate in the study, your data may be sent outside of the Cleveland Clinic for additional analysis and development of the assessment tool used in this study, provided, however, that personal information that could identify you will be removed before data is shared. The research done with your data may lead to the development of new products. You will not receive, either now or in the future, any compensation, royalty, or other financial benefits resulting from any product, procedure, or other items developed from studying your data.

#### What Happens to the Research Equipment at the End of the My Participation?

At the conclusion of your research participation, the bicycle you used (if applicable) will be collected by a contracting company scheduled by research personnel. You will not be financially responsible for any costs associated with the bicycle, its delivery, or its pick-up at the end of the study. Bicycles may be utilized by future participants in the study, and are not available for private purchase. All research participants may keep their Garmin activity monitor.

#### **ALTERNATIVES**

This study is being performed for research purposes only. The alternative to study participation is simply NOT to participate in the investigation.

## **RISKS**

What are the risks of participating in the research study?

#### Cardiac Risks

There are cardiac risks associated with participating in intensive exercise training. Although very rare, during exercise you may experience a serious cardiac (affecting your heart) event. An

example of a cardiac event would be a heart attack or another medical condition that causes damage to your heart or cardiovascular system. Potential symptoms of a cardiac event may include any of the following: chest tightness or pressure, difficulty catching your breath, dizziness or fainting, fatigue, fluid buildup, your heart pounding or racing, pain or numbness in your arms or legs, and/or abdominal pain, nausea or vomiting. If you experience any of these symptoms while completing unsupervised exercise, seek emergency treatment immediately, as these types of symptoms may be related to a cardiac event, and can be fatal.

#### Feeling of discomfort off of Parkinson's disease medications:

Withholding your Parkinson's disease medications may be uncomfortable for you. You may experience an increase in your Parkinson's disease symptoms off-medications (i.e. increased tremors, increased rigidity, slowness of movement, or generalized discomfort).

## Feelings of loss of balance or dizziness:

The testing involves a series of balance assessments that may cause you to experience a feeling of dizziness, headache, nausea, or a general sense of fogginess. You may discontinue the testing at any time. This risk may be higher, and you may feel dizzier during your "off-medication" appointment. However, a trained research clinician will be standing next to you as a spotter throughout all of the testing.

#### Skin irritation or inflammation (Exercise Group Only):

Skin around your heart rate monitor or in other locations may become irritated during exercise sessions- please move the heart rate monitor to a different area as necessary. Also wear appropriate exercise clothing to help minimize the risk of chafing during exercise.

#### Confidentiality of Data:

Cleveland Clinic and the University of Utah: This is a multi-site study involving the Cleveland Clinic and the University of Utah. Your research participation data will be de-identified prior to sharing information between sites. This means items that can identify you will be replaced with a study number, and only data points will be shared.

- Garmin Activity Tracker: The data from your physical activity monitor that you will be
  asked to wear is managed by Garmin, and will be visible to research study staff at the
  Cleveland Clinic or the University of Utah. A study number will link your information to
  research personnel, and will not be listed on Garmin's on-line portal.
- Peloton Bicycle (Exercisers Only): Peloton (a manufacturer of indoor cycling equipment)
  will maintain your exercise specific data on a portal that will have your study number
  on it. Research study staff at the Cleveland Clinic and the University of Utah will have
  access to your exercise data as part of the study.


#### BENEFITS

You may or may not benefit from participating in this study. Taking part in this study will help researchers learn the impact of an exercise program on the symptoms of Parkinson's disease.

## **COSTS**

#### Are there any costs to you if you participate in this study?

As part of your study participation, you will be screened via telephone for your safety in an exercise study using the American College of Sports Medicine questionnaire. If you need additional clearance from your doctor, you will be responsible for obtaining that letter. If an appointment is required, you will be responsible for any costs associated with that appointment. You will need Wi-Fi and a smartphone to participate in this study. If you choose to participate, but do not currently have one or both of these technologies, you will need to purchase them at your own expense.

### **PAYMENTS**

### Are there any payments to you if you participate in this study?

You will receive a \$50.00 check issued to you by the Cleveland Clinic for each assessment you complete, for a possible total of \$250.00. The check will be mailed to your home address.

Your social security number is only required for compensation. You may choose to participate in the study without compensation if you chose not to disclose your social security number.

The IRS requires the Cleveland Clinic Foundation to report payments to an individual of \$600.00 or greater (in a calendar year) on a Form 1099-MISC. Your name, address and social security number will be collected to track the payments made to you, and if you receive \$600.00 or greater, will be used to process a 1099-MISC.

## CONFIDENTIALITY

## What will happen to your information that is collected for this research?

Your study information will be shared, without anyone knowing that it is related to you specifically, with others or use it to research projects not listed in this form. Your data may be stored and shared for future research without additional informed consent if identifiable private information, such as your name and medical record number, are removed. If your identifying information is removed from your data, we will no longer be able to identify and destroy them.

Study results may be shared in medical journals, at scientific meetings, and in other mediums without your identifying information. Your records will be confidential and your identity will not be shared in medical journals, at scientific meetings, and in other mediums without your express consent.

To further protect your privacy, we have obtained a Certificate of Confidentiality from the United States Department of Health and human Services (DHHS) and the National Institutes of Health (NIH). With this Certificate, we cannot be forced (for example by court order or subpoena) to disclose information that may identify you in any federal, state, local, civil, criminal, legislative, administrative, or other proceedings. The researchers will use the Certificate to resist demands for information that would identify you except to prevent serious harm to you or others, and as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). No voluntary disclosure of your information will be made.

You should understand that a Certificate of Confidentiality does not prevent you, or a member of your family, from voluntarily releasing information about yourself or your involvement in this research. If an insurer or employer learns about your participation, and obtains your consent to receive research information, then we may not use the Certificate of Confidentiality to withhold this information. This means that you and your family must also actively protect your own privacy.

#### **Clinical Trials Registry**

A description of this clinical trial will be available at <a href="https://clinicaltrials.gov">https://clinicaltrials.gov</a>, as required by U. S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search the website at any time.


## **QUESTIONS**

## Who do you call if you have any questions or problems?

If you have any questions about the research or develop a research-related problem, you should contact the Principal Investigator or the study coordinator at your site. If you have questions about your rights as a research subject, you should contact the Cleveland Clinic Institutional Review Board at (216) 444-2924.

## **VOLUNTARY PARTICIPATION**

## What are your rights as a research participant?

Taking part in this study is voluntary. You will be told of any new, relevant information from the research that may affect your health, welfare, or willingness to continue in this study. You may choose not to take part or may leave the study at any time. Withdrawing from the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to withdraw from the study you should discuss with your study doctor your decision to ensure a safe withdrawal.

You are free to withdraw consent at any time and to discontinue participation in the research study. Such discontinuation will not affect your regular treatment or medical care in any way. If you wish to withdraw, you should notify the Principal Investigator that you no longer want to participate in this study. In addition, your study doctor may decide to end your participation in this study at any time after he has explained the reasons for doing so and has helped arrange for your continued care by your own doctor, if needed.

## PART 2: LOCAL SITE INFORMATION

## SITE NAME

#### **Cleveland Clinic**

## SITE PRINCIPAL INVESTIGATOR

Dr. Jay Alberts 9500 Euclid Ave., ND20 Cleveland, OH 44195 216-445-3222

## CONTACT INFORMATION

Who do you contact with questions about the study?

If you have any questions, you can ask the Site Investigator, (see information above) and/or research staff Elizabeth Jansen at 216-445-3866.

Who do you contact after hours or in case of an emergency?

If you need to contact study staff outside normal business hours, you may contact Dr. Jay Alberts at 440-708-3735.

Where can you get more information?

If the researchers cannot be reached, or if you would like to talk to someone other than the researcher(s) about concerns regarding the study, research participant's rights, research-related injury, or other human subjects research issues, you may contact the Cleveland Clinic Institutional Review Board at (216) 444-2924.

## RESEARCH RELATED INJURY

What will happen if you are injured as a result of taking part in the research? In the event you suffer a research related injury as a result of being in this study, the costs for medical treatment may be billed to you or your medical insurance plan, if applicable. Medical

insurance plans may or may not cover costs for medical treatment of research-related injuries. If you have insurance, you should check with your medical insurance plan before deciding to participate in this research study. In the event your medical insurance plan covers some or all of the treatment costs, you may still be responsible for co-pays or deductibles as required by your medical insurance plan.

Cleveland Clinic has not set aside any money to pay you or to pay for your treatment if you suffer a research related injury as a result of being in the study. There are no plans for Cleveland Clinic to provide other forms of compensation (such as lost wages, pain and suffering, or other direct or indirect losses) to you for research related injuries. You are not waiving any legal rights by signing this form, including the right to seek compensation for an injury.

## HIPAA AUTHORIZATION

#### **HIPAA AUTHORIZATION**

# Authorization to Use or Disclose (Release) Health Information that Identifies You for a Research Study

If you volunteer to participate in this research, you are permitting your site, the Principal Investigator, and the research staff to create, collect, use, store, and share protected health information (PHI) that identifies you for the purposes of this research.

The PHI that we may use or disclose (release) for this research may include your name, address, phone number, date of birth, Social Security number, information from your medical record, lab tests, or certain information relating to your health or condition.

Some of the tests and procedures done solely for this research study may also be placed in your medical record so other doctors know you are in this study. Upon completion of the study, you may have access to the research information that is contained in your medical record.

In addition to the investigators and research staff, your PHI may be looked at by other groups involved with the study such as the Institutional Review Board. Your PHI may also be used by and/or disclosed (released) to:

- Each other and with other researchers involved with the study;
- Law enforcement or other agencies, when required by law;
- The sponsor/funding agency of the research, Garmin (a company that measures your physical activity, accessible through an on-line portal), Peloton Indoor Cycle (a company that manufactures stationary bicycles, and measures, collects, and displays your exercise specifics through an on-line portal) as required to conduct the research and/or confirm the results of the research;
- Non-Cleveland Clinic collaborators of the research study: University of Utah; and

With representatives of government agencies (e.g., Food and Drug Administration, The
Department of Health and Human Services, etc.), review boards including the Cleveland
Clinic Institutional Review Board and its representatives, and other persons who watch over
the conduct of research (e.g., data safety and monitoring boards).

Once your personal health information is released it may be re-disclosed and no longer protected by privacy laws.

Through your use of the Garmin and/or Peloton platforms, applications and service (collectively "Platform") your personal information may be shared with Garmin, Peloton and their partners, including information that you may directly provide, such as your name, email address, telephone number, date of birth, gender, personal health information, device information, message preferences, IP (Internet Protocol) address and other identifiable information. Garmin, Peloton and/or their partners may also collect information from their Platforms by automated means, such as cookies, web server logs, pixel tags/web beacons, and similar technologies which may be used for the provider's advertising networks, analysis services, and/or to improve the function. Information submitted through the Platform(s) may be stored and used by Garmin, Peloton and/or their partners even after the end of the study. You should carefully consider what information you make available through said Platform(s) and carefully review and consider Garmin and Peloton's Terms of Use and Privacy Policies before providing information through said Platform(s).

Your research information may be used and disclosed indefinitely, but you may stop these uses and disclosures at any time by writing to the **Site Principal Investigator** (see first page of Part 2).

Your participation in the research will stop, but any information previously recorded about you cannot be removed from the records and will continue to be used as part of this research. Also, information already disclosed outside your site cannot be retrieved. This will not affect your rights to treatment or benefits outside the research study.

Your site will not use your information collected in this study for another research purpose without your written permission; unless an Institutional Review Board assures your privacy and confidentiality is protected. The IRB is a committee whose job it is to protect the safety and welfare of research subjects.

By signing this informed consent form, you are authorizing such access to your research and medical record information. If you choose not to sign this consent form, you will not be able to participate in this research study. This Authorization does not have an expiration date.


Signature of person obtaining consent

## **SIGNATURES**

Statement of the Participant

I have read and have had verbally explained to me the above information and have had all my questions answered to my satisfaction. I understand that my participation is voluntary and that I may stop my participation in the study at any time. Signing this form does not waive any of my legal rights. I understand that a copy of this consent will be provided to me. By signing below, I agree to take part in this research study.

Printed name of Participant

Date

Statement of the Person Conducting Informed Consent Discussion

I have discussed the information contained in this document with the participant and it is my opinion that the participant understands the risks, benefits, alternatives and procedures involved with this research study.

Printed name of person obtaining consent

Date